CLINICAL TRIAL: NCT06797076
Title: Evaluating an App-Based Treatment for Migraine: The Health enSuite Migraine Study
Brief Title: App-Based Migraine Treatment: The Health enSuite Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Patrick J. McGrath, Principal Investigator, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1031367; 1018439 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura
Keywords: Headache; Migraine; Cognitive Behavioral Therapy
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura; Headache

STUDY DESIGN:
Intervention Model Description: This project consists of a pragmatic randomized controlled trial (RCT). The Consolidated Standards of Reporting Trials (CONSORT) recommendations (http://www.consort-statement.org/) will guide the methodology. Participants will be randomly allocated in a 1:1 ratio to either the intervention group or a waitlist control group. Participants in both groups will complete self-assessments including key outcome measures at baseline before starting the study, at two months post-randomization, and again at six months post-randomization. Participants in the intervention group will receive the full Health enSuite Migraine program described below immediately after being randomized to this group. Participants in the waitlist control group will be waitlisted during the study. After their participation in the study has ended, participants in the waitlist control group will be given access to the full Health enSuite Migraine program for two months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Health enSuite: Migraine has been designed based on established cognitive-behavioral treatments for migraine headache and adapted to fit an automated interactive platform available via an internet-enabled device. The program is divided into a series of treatment modules that will be delivered over 8 weeks. The online program combines treatment elements that are effective in preventing and managing migraine headache pain, including trigger management, stress management, relaxation techniques, cognitive reappraisal, and psychoeducation.
  Interventions: Behavioral: Health enSuite Headache
- Waitlist Control (No Intervention): Participants allocated to the control group will not receive Health enSuite Migraine until after their participation in the trial has ended. During the trial, they will receive treatment as usual and will not be restricted from accessing other standard care services for migraine headache treatment.

INTERVENTIONS:
Behavioral: Health enSuite Headache — The program consists of treatment modules delivered over 8 weeks. Modules include topics such as Headaches and Triggers, Relaxation, Breathing, Changing Thoughts, Imagery, Problem Solving, Nutrition, Sleep, Exercise, Medication, and more. Each module features sections like Goals, Getting Started, Let's Talk, and a Quiz, with Let's Practice in four modules. Intervention participants track headaches using a structured tracker to log impacts, daily events (e.g., exposure, strategies, medication), and notes. Control group participants track headaches only at baseline, two months, and five months post-randomization. Weekly reminders ("nudges") encourage app usage, with the same frequency for all users. Reports summarizing daily headache data are available to participants.
  Arms: Intervention

SUMMARY:
Health enSuite is a suite of applications designed by our research team at the Centre of Research in Family Health at IWK Health. These applications evaluate virtual solutions for clinical problems and assist family doctors with their adult patients.

Health enSuite will be utilized by Canadian family physicians targeting insomnia, anxiety, migraine headache, and caregiver distress.

Health enSuite Migraine has been designed to make cognitive and behavioral techniques for managing migraine headache readily available to primary care patients. The online program combines treatment elements that are effective in preventing and managing migraine headache pain, including trigger management, stress management, relaxation techniques, cognitive reappraisal, and psychoeducation.

DETAILED DESCRIPTION:
Headaches are highly prevalent among Canadians and many people visit their primary care provider due to headache symptoms. Headaches can be classified based on frequency (acute, episodic, chronic) and symptom presentation (migraine headache, tension-type, cluster, etc.). Headaches are of concern to many people as the World Health Organization (WHO) has reported that in 2016, more than half of people around the world between 16-65 years old reported having headaches. Up to 70% of individuals experience tension headaches, and 8.3% of Canadians are affected by migraine headache.

Headache symptoms can last a few hours to several days and are debilitating as they cause significant pain and distress. Headaches can also negatively impact one's life as they cause problems related to work performance and/or school activities (i.e., not being able to complete an assignment or project on time).

People who seek medical attention from their primary care provider for their headache pain often have difficulty receiving adequate treatment. One of the barriers to the optimal treatment of headaches is that the availability of non-pharmacological, psychosocial treatments is very limited. Although medications can be an important part of effective headache management, the use of non-pharmacological treatments is widely recommended .

Among headache disorders, migraine headaches are particularly debilitating due to their neurological basis, severity, and high burden on daily functioning. Unlike tension-type headaches, migraine headaches involve additional symptoms such as nausea, photophobia, and phonophobia, leading to greater disability. Given this significant impact, our study focuses specifically on developing a digital Cognitive Behavioral Therapy (CBT) intervention for migraine headache sufferers.

The National Canadian Migraine Strategy has recommended self-management patient interventions and patient education to learn skills to manage their symptoms in partnership with their healthcare providers. They have also advocated for the use of non-pharmacological therapies like stress management, skills to avoid triggers causing migraine headache, relaxation therapies, and self-monitoring for the management of migraine headache as part of their chronic disease management program for migraine headache. Although many medications can reduce pain due to migraine headache, their frequent use has associated side effects, and the prolonged use or overuse of medications can also cause migraine headache. Thus, an overreliance on pharmacological treatments and a lack of attention to lifestyle and psychosocial factors contributing to migraine headache symptoms can create sub-optimal outcomes for patients. Therefore, our goal is to develop a CBT program for migraine headache that can be delivered through an internet-connected phone, tablet, or computer and provide effective treatment to a wide range of patients with migraine headache. Health enSuite is a suite of applications designed by our research team at the Centre of Research in Family Health at IWK Health. Health enSuite will be utilized by patients suffering from insomnia, anxiety, migraine headache, and caregiver distress.

Health enSuite Migraine has been designed to make cognitive and behavioral techniques for managing migraine headache readily available to people suffering from migraine headache. The online program combines treatment elements that are effective in preventing and managing migraine headache pain, including trigger management, stress management, relaxation techniques, cognitive reappraisal, and psychoeducation.

ELIGIBILITY:
Inclusion Criteria (for study entry):

* Fluent in English
* Age 18 to 50 years
* Regular access to an internet-connected device (e.g., smartphone, tablet, or computer)
* Scores 2 or more on the ID Migraine Screener

Inclusion Criteria (for enrollment):

* Completes at least 50% of the daily entries when asked to use the migraine headache tracker for a 28-day period
* Experiences migraine headache on at least 4 days, but no more than 20 days, within the past month (based on diary data)

Exclusion Criteria:

* Diagnosis of psychosis and/or schizophrenia
* Physical or cognitive impairment that compromises ability to provide informed consent
* Pregnancy, planning pregnancy during the study, or currently breastfeeding
* Change in medications and/or dietary supplements (herbal supplements, minerals, vitamins) for migraine headache pain in the past month

Rationale for Eligibility Criteria:

Behavioural and/or psychosocial treatment is not recommended for migraine headache related to conditions such as psychosis, and/or schizophrenia. While behavioral and psychosocial treatments may offer some benefits for individuals with migraine headache related to psychosis and schizophrenia, there are also potential risks to consider. For example, CBT may involve exploring painful feelings and experiences, which could be distressing for individuals with psychosis. This could potentially exacerbate psychotic symptoms or lead to emotional distress. Additionally, some individuals with schizophrenia may have difficulty engaging in CBT due to cognitive impairments, such as difficulty concentrating or remembering information, or paranoia. Therefore, potential participants who have any of these conditions will be excluded from the study.

Pregnancy and breastfeeding result in hormonal changes that can increase migraine headache symptoms. Thus, guidelines for headache trials highly suggest excluding participants who are planning to be pregnant, currently pregnant or are nursing their infants.

The initiation of other treatments for migraine headache at the same time as Health enSuite Migraine could jeopardize the interpretation of the trial results. They are permitted to continue using any pre-existing treatments (medications, dietary supplements, vitamins). If participants are taking any medications/ and or dietary supplements, they must have been taking them for at least one month to be eligible for enrollment in the trial. Participants are asked at the end of the trial if they have started any new medication while using Health enSuite Migraine; if the new medication taken is recognized to have impacted the results, the participant's data will be removed for data analysis.

The age range of 18-50 years was chosen to align with the typical demographic most affected by migraine headache and to ensure the app's design and content are appropriate for its intended users. Research indicates that migraine headaches are most prevalent in this age group, with peak incidence occurring during early adulthood and middle age. Additionally, individuals outside this range, such as adolescents or older adults, may have distinct physiological, psychological, and treatment needs that differ from those of the target demographic.

For example, older adults often experience migraine headache differently due to age-related comorbidities or medication interactions, which may require specialized interventions beyond the scope of this study or app. Similarly, the app's features and usability are tailored to adults with regular access to technology and familiarity with app-based interventions.

The Health enSuite Migraine program being tested in this trial requires the use of an internet-connected device. Health enSuite Migraine can be accessed through the web browser on an electronic device with an internet connection. People who do not have regular access to an internet-connected device are unlikely to benefit from Health enSuite Migraine, and therefore they will be excluded.

Participants must have experienced migraine headache pain at least four days out of each month. This criterion is intended to ensure that all participants will experience at least some migraine headache symptoms throughout the study. Chronic daily migraine headaches are especially difficult to treat through psychosocial intervention alone, therefore participants who report migraine headache on more than 20 days per month will be excluded. Apart from the above mentioned 8 criteria points, study eligibility will be evaluated based on one month of daily migraine headache tracking completed at baseline to ensure the participant experiences a migraine headache between 4 to 20 days within the past month

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 415 (Estimated)
Dates: Start 2026-02-15 (Estimated); Primary Completion 2027-01-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Change in Migraine Headache Frequency | Baseline assessment, 2 months post randomization, 5 months post randomization
  Migraine headache frequency will be tracked using the electronic migraine headache tracker within the Health enSuite Migraine app. The outcome is the change from baseline in the number of migraine headache days.
  Unit of Measure: Number of migraine headache days per month

SECONDARY OUTCOMES:
Responder Rate for Migraine Headache | Baseline assessment, 2 months post randomization, 5 months post randomization
  Percentage of participants achieving ≥30% reduction in migraine headache days from baseline, measured via the migraine headache tracker.
  Unit of Measure: % of participants with ≥30% reduction in headache days.
Change in Maximum Migraine Headache Intensity | Baseline assessment, 2 months post randomization, 5 months post randomization
  Maximum headache intensity will be self-reported using the migraine headache tracker.
  Unit of Measure: Intensity score (0-10 scale)
Change in Migraine-Related Functional Impairment (MIDAS) | Baseline assessment, 2 months post randomization, 5 months post randomization
  The Migraine Disability Assessment (MIDAS) questionnaire will be used to measure functional impairment due to migraine. The outcome is the change in MIDAS total score.
  Unit of Measure: MIDAS total score (0-21+)
Change in Depression Symptoms (PHQ-9) | Baseline assessment, 2 months post randomization, 5 months post randomization
  Depression symptoms will be measured using the 9-item Patient Health Questionnaire (PHQ-9). The outcome is the change in PHQ-9 total score.
  Unit of Measure: PHQ-9 total score (0-27)
Changes in Daily Factors Related to Migraine Episodes | Baseline assessment, 2 months post randomization, 5 months post randomization
  Exploratory assessment of daily self-reported factors (sleep, mood, emotional state, environmental exposures, dietary intake, coping strategies, and medication use) and their association with migraine episodes, as reported in the optional components of the migraine headache tracker.
  Unit of Measure: Self-reported diary entries (descriptive/exploratory; no single standardized unit)
Changes from baseline in daily factors | Baseline assessment, 2 months post randomization, 5 months post randomization
  such as sleep, mood, emotional state, environmental exposures, dietary intake, coping strategies, and medication use, and their potential associations with migraine episodes, as self-reported in the optional components of the migraine headache tracker.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Patrick, Principal Investigator — IWK Health Centre

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets may be retained and stored within the Centre for Research in Family Health as required for future research or program development, if merited. During Consent, participants will be offered the option of allowing their de-identified study data to be re-used by other approved researchers under the conditions that the research projects are approved by an appropriate ethics board and the researchers sign an agreement ensuring confidentiality and restricting data use only to the approved study. A database will be created containing only the data for those participants who agree will be available to researchers who meet these criteria.
Time Frame: From study closure to five years post publication.
Access Criteria: During Consent, participants will be offered the option of allowing their de-identified study data to be re-used by other approved researchers under the conditions that the research projects are approved by an appropriate ethics board and the researchers sign an agreement ensuring confidentiality and restricting data use only to the approved study.

REFERENCES:
- [Background] Becker WJ. Weather and migraine: can so many patients be wrong? Cephalalgia. 2011 Mar;31(4):387-90. doi: 10.1177/0333102410385583. Epub 2010 Dec 16. No abstract available. PMID 21163817
- [Background] Lipton RB, Stewart WF, Sawyer J, Edmeads JG. Clinical utility of an instrument assessing migraine disability: the Migraine Disability Assessment (MIDAS) questionnaire. Headache. 2001 Oct;41(9):854-61. PMID 11703471
- [Background] World Health Organization. (2016). World Health Statistics 2016 [OP]: Monitoring Health for the Sustainable Development Goals (SDGs). World Health Organization.
- [Background] Ramage-Morin PL, Gilmour H. Prevalence of migraine in the Canadian household population. Health Rep. 2014 Jun;25(6):10-6. PMID 24941316
- [Background] Becker WJ. Cervicogenic headache: evidence that the neck is a pain generator. Headache. 2010 Apr;50(4):699-705. doi: 10.1111/j.1526-4610.2010.01648.x. PMID 20456156
- [Background] Lipton RB, Bigal ME, Kolodner K, Stewart WF, Liberman JN, Steiner TJ. The family impact of migraine: population-based studies in the USA and UK. Cephalalgia. 2003 Jul;23(6):429-40. doi: 10.1046/j.1468-2982.2003.00543.x. PMID 12807522
- [Background] Abu Bakar N, Tanprawate S, Lambru G, Torkamani M, Jahanshahi M, Matharu M. Quality of life in primary headache disorders: A review. Cephalalgia. 2016 Jan;36(1):67-91. doi: 10.1177/0333102415580099. Epub 2015 Apr 17. PMID 25888584
- [Background] Lipton RB, Hamelsky SW, Kolodner KB, Steiner TJ, Stewart WF. Migraine, quality of life, and depression: a population-based case-control study. Neurology. 2000 Sep 12;55(5):629-35. doi: 10.1212/wnl.55.5.629. PMID 10980724
- [Background] Linde M, Jonsson P, Hedenrud T. Influence of disease features on adherence to prophylactic migraine medication. Acta Neurol Scand. 2008 Dec;118(6):367-72. doi: 10.1111/j.1600-0404.2008.01042.x. Epub 2008 May 27. PMID 18513346
- [Background] Lipton RB, Bigal ME, Diamond M, Freitag F, Reed ML, Stewart WF; AMPP Advisory Group. Migraine prevalence, disease burden, and the need for preventive therapy. Neurology. 2007 Jan 30;68(5):343-9. doi: 10.1212/01.wnl.0000252808.97649.21. PMID 17261680
- [Background] Dodick DW, Loder EW, Manack Adams A, Buse DC, Fanning KM, Reed ML, Lipton RB. Assessing Barriers to Chronic Migraine Consultation, Diagnosis, and Treatment: Results From the Chronic Migraine Epidemiology and Outcomes (CaMEO) Study. Headache. 2016 May;56(5):821-834. doi: 10.1111/head.12774. Epub 2016 May 3. PMID 27143127
- [Background] Becker WJ, Findlay T, Moga C, Scott NA, Harstall C, Taenzer P. Guideline for primary care management of headache in adults. Can Fam Physician. 2015 Aug;61(8):670-9. PMID 26273080
- [Background] Diener HC, Dodick D, Evers S, Holle D, Jensen RH, Lipton RB, Porreca F, Silberstein S, Schwedt T. Pathophysiology, prevention, and treatment of medication overuse headache. Lancet Neurol. 2019 Sep;18(9):891-902. doi: 10.1016/S1474-4422(19)30146-2. Epub 2019 Jun 4. PMID 31174999
- [Background] Penzien DB, Andrasik F, Freidenberg BM, Houle TT, Lake AE 3rd, Lipchik GL, Holroyd KA, Lipton RB, McCrory DC, Nash JM, Nicholson RA, Powers SW, Rains JC, Wittrock DA; American Headache Society Behavioral Clinical Trials Workgroup. Guidelines for trials of behavioral treatments for recurrent headache, first edition: American Headache Society Behavioral Clinical Trials Workgroup. Headache. 2005 May;45 Suppl 2:S110-32. doi: 10.1111/j.1526-4610.2005.4502004.x. PMID 15921503
- [Background] Whyte CA, Tepper SJ. Adverse effects of medications commonly used in the treatment of migraine. Expert Rev Neurother. 2009 Sep;9(9):1379-91. doi: 10.1586/ern.09.47. PMID 19769452
- [Background] Tepper SJ. Medication-overuse headache. Continuum (Minneap Minn). 2012 Aug;18(4):807-22. doi: 10.1212/01.CON.0000418644.32032.7b. PMID 22868543
- [Background] Bromberg J, Wood ME, Black RA, Surette DA, Zacharoff KL, Chiauzzi EJ. A randomized trial of a web-based intervention to improve migraine self-management and coping. Headache. 2012 Feb;52(2):244-61. doi: 10.1111/j.1526-4610.2011.02031.x. PMID 22413151
- [Background] Devineni T, Blanchard EB. A randomized controlled trial of an internet-based treatment for chronic headache. Behav Res Ther. 2005 Mar;43(3):277-92. doi: 10.1016/j.brat.2004.01.008. PMID 15680926
- [Background] Hedborg K, Muhr C. Multimodal behavioral treatment of migraine: an Internet-administered, randomized, controlled trial. Ups J Med Sci. 2011 Aug;116(3):169-86. doi: 10.3109/03009734.2011.575963. Epub 2011 Apr 20. PMID 21506633
- [Background] Strom L, Pettersson R, Andersson G. A controlled trial of self-help treatment of recurrent headache conducted via the Internet. J Consult Clin Psychol. 2000 Aug;68(4):722-7. PMID 10965647
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Bae JY, Sung HK, Kwon NY, Go HY, Kim TJ, Shin SM, Lee S. Cognitive Behavioral Therapy for Migraine Headache: A Systematic Review and Meta-Analysis. Medicina (Kaunas). 2021 Dec 28;58(1):44. doi: 10.3390/medicina58010044. PMID 35056352
- [Background] Koh, K. (2018). Cognitive behavioral therapy for patients with chronic headache: Biopsychosociospiritual perspectives. In Handbook of behavioral medicine (pp. 269-277). Springer. https://doi.org/10.1007/978-3-030-02783-4_18
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. The Patient Health Questionnaire Somatic, Anxiety, and Depressive Symptom Scales: a systematic review. Gen Hosp Psychiatry. 2010 Jul-Aug;32(4):345-59. doi: 10.1016/j.genhosppsych.2010.03.006. Epub 2010 May 7. PMID 20633738
- [Background] Mitchell AJ, Yadegarfar M, Gill J, Stubbs B. Case finding and screening clinical utility of the Patient Health Questionnaire (PHQ-9 and PHQ-2) for depression in primary care: a diagnostic meta-analysis of 40 studies. BJPsych Open. 2016 Mar 9;2(2):127-138. doi: 10.1192/bjpo.bp.115.001685. eCollection 2016 Mar. PMID 27703765
- [Background] Kroenke K. Enhancing the clinical utility of depression screening. CMAJ. 2012 Feb 21;184(3):281-2. doi: 10.1503/cmaj.112004. Epub 2012 Jan 9. No abstract available. PMID 22231681
- [Background] British Columbia Medical Association. (2002). Guidelines and Protocols Advisory Committe. Acute otitis media (AOM).
- [Background] Titov N, Andrews G, Davies M, McIntyre K, Robinson E, Solley K. Internet treatment for depression: a randomized controlled trial comparing clinician vs. technician assistance. PLoS One. 2010 Jun 8;5(6):e10939. doi: 10.1371/journal.pone.0010939. PMID 20544030
- [Background] Richards DA, Lovell K, Gilbody S, Gask L, Torgerson D, Barkham M, Bland M, Bower P, Lankshear AJ, Simpson A, Fletcher J, Escott D, Hennessy S, Richardson R. Collaborative care for depression in UK primary care: a randomized controlled trial. Psychol Med. 2008 Feb;38(2):279-87. doi: 10.1017/S0033291707001365. Epub 2007 Sep 6. PMID 17803837
- [Background] Gilbody S, Richards D, Barkham M. Diagnosing depression in primary care using self-completed instruments: UK validation of PHQ-9 and CORE-OM. Br J Gen Pract. 2007 Aug;57(541):650-2. PMID 17688760
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Eilert N, Enrique A, Wogan R, Mooney O, Timulak L, Richards D. The effectiveness of Internet-delivered treatment for generalized anxiety disorder: An updated systematic review and meta-analysis. Depress Anxiety. 2021 Feb;38(2):196-219. doi: 10.1002/da.23115. Epub 2020 Nov 22. PMID 33225589
- [Background] Stewart WF, Lipton RB, Dowson AJ, Sawyer J. Development and testing of the Migraine Disability Assessment (MIDAS) Questionnaire to assess headache-related disability. Neurology. 2001;56(6 Suppl 1):S20-8. doi: 10.1212/wnl.56.suppl_1.s20. PMID 11294956
- [Background] Dowson, A., Salt, R., & Kilminster, S. (2004). The outcome of headache management following nurse intervention: Assessment in clinical practice using the Migraine Disability Assessment (MIDAS) questionnaire. Headache Care, 1, 177-181. https://doi.org/10.1185/174234304125004532
- [Background] Edmeads J, Lainez JM, Brandes JL, Schoenen J, Freitag F. Potential of the Migraine Disability Assessment (MIDAS) Questionnaire as a public health initiative and in clinical practice. Neurology. 2001;56(6 Suppl 1):S29-34. doi: 10.1212/wnl.56.suppl_1.s29. PMID 11294957
- [Background] Kelman L. Migraine changes with age: IMPACT on migraine classification. Headache. 2006 Jul-Aug;46(7):1161-71. doi: 10.1111/j.1526-4610.2006.00444.x. PMID 16866720
- [Background] Lipton RB, Scher AI, Kolodner K, Liberman J, Steiner TJ, Stewart WF. Migraine in the United States: epidemiology and patterns of health care use. Neurology. 2002 Mar 26;58(6):885-94. doi: 10.1212/wnl.58.6.885. PMID 11914403
- [Background] Onan D, Younis S, Wellsgatnik WD, Farham F, Andruskevicius S, Abashidze A, Jusupova A, Romanenko Y, Grosu O, Moldokulova MZ, Mursalova U, Saidkhodjaeva S, Martelletti P, Ashina S. Debate: differences and similarities between tension-type headache and migraine. J Headache Pain. 2023 Jul 21;24(1):92. doi: 10.1186/s10194-023-01614-0. PMID 37474899